CLINICAL TRIAL: NCT04295720
Title: Treatment of Post-Chemotherapy Cognitive Impairment With Transcranial Magnetic Stimulation (Chemobrain TMS)
Brief Title: Treatment of Post-Chemo Cognitive Impairment w/Transcranial Magnetic Stimulation (Chemobrain TMS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Stopped due to the risk of COVID-19 variants to our subject base of cancer patients
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1911180572
Record Dates: First submitted 2020-02-27; First posted 2020-03-04 (Actual); Results first posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Chemo-brain
Keywords: Chemo-brain; Post-Chemotherapy cognitive impairment; PCCI; Transcranial magnetic stimulation; TMS
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: 12 participants with PCCI will be recruited to participate in this trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Transcranial magnetic stimulation (TMS) (Experimental): We propose to test the efficacy of rTMS for the treatment of PCCI. Efficacy measures will include baseline and post-rTMS neuropsychological testing, functional MRI and biometry data using body worn sensors.
  Interventions: Device: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: Transcranial magnetic stimulation (TMS) — Subjects will undergo testing at baseline prior to TMS treatments and once more at the end of the 2-week intervention.After the conclusion of baseline data acquisition, the research team will analyze each participant's unique structural and functional connectivity patterns to determine stimulation site for TMS in future study sessions.
  The subjects will receive 10-sessions (1 session per day, M-F over 2 consecutive weeks).
  The treatment itself lasts approximately only 190 seconds.

SUMMARY:
In this pilot study, the investigators propose to test the efficacy of rTMS for the treatment of PCCI. Efficacy measures will include baseline and post-rTMS neuropsychological testing, functional MRI and biometry data using body worn sensors.

DETAILED DESCRIPTION:
Transcranial magnetic stimulation (TMS) is a safe and non-invasive brain stimulation technique. It uses a magnetic coil to stimulate brain tissue painlessly using only a magnet (no electrodes or electrical wires) in a procedure that does not involve any surgery or sedation. TMS is currently FDA approved to treat depression and migraines. Although this technology is applicable to many other brain conditions as well, it has not been systematically examined in individuals with "Chemo-brain". Chemo-brain or Post-Chemotherapy Cognitive Impairment (PCCI) is defined as cognitive changes including impairment of memory, learning, concentration, reasoning, executive function, attention and visuo visio-spatial skills that occur during or after chemotherapy treatment.

In this study, investigators will:

1. use high-resolution magnetic resonance imaging (MRI) of individuals' brains to determine precisely where to place the TMS magnetic coil in order to stimulate the target brain region based off their unique brain structure.
2. use TMS to stimulate the target region of the brain.
3. take high-resolution MRI pictures of the brain both baseline and post-TMS to study whether the brain activity of the target region changes as a result of the TMS stimulation.
4. perform neuropsychological tasks baseline and post-TMS to study if performance is improved following stimulation of the target brain region.
5. collect data from completing Frailty assessments, baseline and post-TMS.
6. study the short-term and long-term treatment effects.
7. collect subject's daily activity and sleep/wake patterns from watch style device (http://www.actigraphy.com/solutions/actiwatch/actiwatch-plus-specifications.html).
8. perform behavioral assessments, baseline and post-TMS, to study whether there are measurable changes following stimulation of the target brain region.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>=18).
* PCCI diagnosis (see information below).
* Right Handed (We will not enroll left-handed dominant people because they tend to have more symmetric brain function and thus targeting the left frontal region may not be as effective.)
* English speaking.
* Cancer treatment completed and considered curative with the exception of endocrine therapy after chemotherapy.
* Able to attend daily intervention (Monday-Friday) for 2 weeks.
* Not enrolled in another interventional study within 6 months prior to beginning this study.

Exclusion Criteria:

* Pregnancy or thinking of becoming pregnant.
* Undergoing active treatment for cancer.
* Routine contraindications for MRI (including incompatible medical implants or metal fragments in the body at risk for migration or heating with application of the magnetic field) including severe claustrophobia.
* History of brain metastasis or other brain tumor.
* History of stroke or traumatic brain injury.
* Frequent or severe headaches.
* Cognitive or mood disorder prior to chemotherapy (i.e. dementia or depression).
* History of epilepsy, or other seizure disorders.
* History mental health disorders, such as substance misuse, bipolar disorder or psychosis.
* Taking medication for seizures or that could lower seizure threshold if withdrawn.
* Inability to complete neuropsychological testing.
* Prior treatment with rTMS. We will enroll subjects without prior experience with rTMS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Kuo, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Magnetic Stimulation (TMS): We propose to test the efficacy of rTMS for the treatment of PCCI. Efficacy measures will include baseline and post-rTMS neuropsychological testing, functional MRI and biometry data using body worn sensors.
  Transcranial magnetic stimulation (TMS): Subjects will undergo testing at baseline prior to TMS treatments and once more at the end of the 2-week intervention.After the conclusion of baseline data acquisition, the research team will analyze each participant's unique structural and functional connectivity patterns to determine stimulation site for TMS in future study sessions.
  The subjects will receive 10-sessions (1 session per day, M-F over 2 consecutive weeks).
  The treatment itself lasts approximately only 190 seconds.
Period: Overall Study
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Transcranial Magnetic Stimulation (TMS): We propose to test the efficacy of rTMS for the treatment of PCCI. Efficacy measures will include baseline and post-rTMS neuropsychological testing, functional MRI and biometry data using body worn sensors.
  Transcranial magnetic stimulation (TMS): Subjects will undergo testing at baseline prior to TMS treatments and once more at the end of the 2-week intervention. After the conclusion of baseline data acquisition, the research team will analyze each participant's unique structural and functional connectivity patterns to determine stimulation site for TMS in future study sessions.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 1
Neuropsychological testing [Mean (Standard Deviation); unit: total number of items recalled correctly] — The Baseline Measure is the combined score of the following Neuropsychological tests prior to the treatment. The score from each test was added together to come up with a single value for comparison with the post treatment assessments.
  A higher score indicates better performance. Minimum is score of 0 and maximum is not applicable (timed test).
  The Neuropsychological tests we analyzed:
  Forward Digit Span Backward Digit Span Rey Auditory Verbal Learning Test Verbal Fluency Task Stroop Color-Word Interference Task
  total number of items recalled correctly | 130 (NA) — Standard Deviation is not calculable for 1 participant

OUTCOME MEASURES:

1. Primary Outcome: Memory Testing
Description: Efficacy measures will include baseline and post-rTMS neuropsychological testing. The Outcome Measure is the difference between the pre and post scores of the following Neuropsychological tests. The score from each test was added together to come up with a single value.
  A higher score indicates better performance. Minimum is score of 0 and maximum is not applicable (a timed test).
  The Neuropsychological tests we analyzed:
  Forward Digit Span Backward Digit Span Rey Auditory Verbal Learning Test Verbal Fluency Task Stroop Color-Word Interference Task
Time Frame: 14 days
Population: 1 participant was analyzed.
Measure: Mean (Standard Deviation); unit: items recalled correctly
Groups:
- Transcranial Magnetic Stimulation (TMS): Efficacy measures will include baseline and post-rTMS neuropsychological testing, functional MRI and biometry data using body worn sensors.
  This is an open label trial with only a treatment arm (no placebo group).
Arm/Group | Transcranial Magnetic Stimulation (TMS)
Number analyzed (Participants) | 1
items recalled correctly | 20 (NA) — Standard Deviation is not calculable for 1 participant

ADVERSE EVENTS:
Time Frame: 14 days
Description: Adverse events were monitored/assessed beginning at initiation of treatment (day 1) through treatment completion, 14 days. Adverse events were monitored by Non-Systematic Assessment method; self-reported by participants.
Arm/Group | Transcranial Magnetic Stimulation (TMS)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT04295720/Prot_SAP_000.pdf